CLINICAL TRIAL: NCT04512547
Title: Oxidative Stress and Regional Airway Remodeling and Fibrosis in Obese Asthma
Brief Title: Oxidative Stress in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00104900
Record Dates: First submitted 2020-07-20; First posted 2020-08-13 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Asthma; Obesity
Keywords: Asthma; MRI; Obesity
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obese Asthmatics (Experimental): Obese patients that come to Duke that have been diagnosed with Asthma will be approached.
  Interventions: Drug: Hyperpolarized 129XeMRI
- Obese Non-Asthmatics (Active Comparator): The obese non-asthmatics will be collected from an IRB pre-approved Healthy Volunteer Data Repository.
  Interventions: Drug: Hyperpolarized 129XeMRI

INTERVENTIONS:
Drug: Hyperpolarized 129XeMRI — Images obtained using 129XeMRI will be obtained on both obese asthmatic and non-asthmatics

SUMMARY:
40% of all asthma patients in the US are obese. Obese asthmatics have more severe disease than lean asthmatics and do not respond as well to conventional anti-inflammatory therapies. This proposal will utilize 3D functional imaging with 129XeMRI and single cell RNA sequencing to study mechanisms driving regional airway remodeling and fibrosis in obese asthma subjects and in preclinical models of obese asthma.

DETAILED DESCRIPTION:
ABSTRACT

Obesity, a major comorbidity and a potential modulator of asthma, affects nearly 40% of asthmatics in the U.S., and increases its severity. Obese asthmatics do not respond as well to conventional anti-inflammatory therapies and new biologics targeting asthma are less effective in obese asthmatics compared to lean. Very little research has been conducted in obese animals or obese asthmatics, resulting in a major knowledge deficit.

A key feature of asthma is airway remodeling and fibrosis, broadly defined as a change in distribution, thickness, composition, mass or volume of structural components of the airway wall of patients relative to healthy patients. Airway remodeling is difficult to diagnose in obese patients as mechanical changes in chest wall compliance can contribute to the physiological changes seen. Classically, evidence of airway remodeling and fibrosis are revealed as fixed airway obstruction on spirometry. However, spirometry is not only insensitive to the peripheral airways, where airway remodeling occurs, but is fundamentally incapable of localizing the sites of remodeling and fibrosis. Thus, a critical research limitation in the study of airway remodeling and fibrosis in asthma is defining regions of disease activity to explore disease-specific mechanisms. To understand the nature of airway remodeling and fibrosis in obese asthma and to rapidly screen for novel therapies requires translation between preclinical models and patients, while using advanced imaging. Recent work in asthma using 3D functional imaging with 129Xe MRI has revealed the location of both reversible and fixed ventilation defects (defined based on bronchodilator responsivity). Several studies suggest that fixed defects represent sites of airway remodeling and fibrosis, but to date, this has been inferred indirectly from sputum analyses and CT scans. The central hypothesis is that sites of abnormal ventilation on 129XeMRI represent areas of airway remodeling and fibrosis and are enriched with fibroblasts that are invasive, proliferative and fibrogenic. It is further hypothesized that regional alterations in oxidant stress driving the production of transforming growth factor-beta (TGF-β) direct pro-remodeling fibroblast functions. Lastly, it is hypothesized that 129XeMRI will be a sensitive and specific biomarker of airway remodeling and fibrosis in obese asthmatics and rat models of obese asthma. By leveraging our excellence in clinical asthma, bronchoscopy, and translational expertise in cell function/signaling and 3D MR imaging in both patients and animal models, both ex vivo cell-specific mechanistic studies and in vivo animal model studies will be conducted to uncover the mechanisms of molecular and cellular function through the following Specific Aims: Aim 1) Identify the pathology, structural cell profile (airway fibroblast and epithelial cell) and redox status corresponding to regional areas of fixed and reversible post-bronchodilator defects (BD) in obese asthmatics; 2) Define the cellular requirement for redox-mediated TGF-β signaling between airway epithelial cells and fibroblasts driving regional remodeling in obese asthma; 3) Develop non-invasive 3D imaging techniques to assess airway regional remodeling in experimental rodent models of obese asthma.

ELIGIBILITY:
Inclusion Criteria:

Asthma Cohort INCLUSION

* Adequate completion of informed consent process with written documentation
* Male and female patients, 18 - 65 years old, inclusive
* Physician diagnosis of asthma for > 1 year
* Able to perform reproducible spirometry according to ATS criteria
* Post-bronchodilator FEV1 ≥ 60% of predicted at Visit 0
* All racial/ethnic backgrounds may participate
* BMI ≥ 30 kg/m2
* Regular treatment with ICS or ICS/LABA and/or LAMA combination medication for at least 3 months; on a stable dose for the 4 weeks prior to Visit 0
* Smoking history <10 pack years and no smoking in the last 3 months
* Late onset asthma: Age of asthma onset (diagnosis) ≥12 years;
* FeNO < 25 ppb at Visit 0
* Negative allergen skin test
* Early onset asthma: Age of asthma onset (diagnosis) <12 years
* FeNO ≥ 25 ppb at Visit 0
* Positive allergen skin test

Non-Asthma Cohort INCLUSION

* No history of asthma or other chronic lung diseases
* Male and female patients, 18 - 65 years old, inclusive
* Not currently smoking or using other forms of tobacco-related products (including vaping)
* Smoking history <10 pack years and no smoking in the past 3 months
* FEV1 > 80% of predicted and FEV1/FVC > lower limit of normal.
* Ability to sign consent
* BMI ≥ 30 kg/m2
* Negative allergen skin test

Additional INCLUSION Criteria for MRI

* Outpatients of either gender, age > 18
* Willing and able to give informed consent and adhere to visit/protocol schedules. (Consent must be given before any study procedures are performed.)
* Women of childbearing potential must have a negative urine pregnancy test prior to MRI.

EXCLUSION Criteria

Asthma Cohort EXCLUSION:

* Respiratory tract infection within the 4 weeks prior to Visit 0
* Oral or systemic corticosteroid burst (for any indication) within the 4 weeks prior to Visit 0. One-time doses, such as intra-articular injections into a shoulder or knee joint, require a 4- week washout prior to Visit 0
* Asthma-related ER visit within the previous 4 weeks of Visit 0
* History of ICU admission/intubation due to asthma in the past 1 year
* Three or more asthma exacerbations requiring treatment with systemic corticosteroids in the past year consistent with severe asthma
* Asthma exacerbation requiring systemic corticosteroids within the 4 weeks prior to Visit 0
* Significant concomitant medical illness, including (but not limited to) heart disease, cancer, uncontrolled diabetes, other chronic lung diseases
* Chronic renal failure (creatinine > 2.0) at Visit 0
* Positive urine pregnancy test at Visit 0 or at any time during the study
* Untreated sleep apnea
* Participation in an intervention study (including, bronchoscopy) or use of investigative drugs within the past 30 days or plans to enroll in such a trial during the study
* Unable or unlikely to complete study assessments in the opinion of the Investigator
* Study intervention poses undue risk to patient in the opinion of the Investigator
* History of bronchial thermoplasty

Non-Asthma Cohort EXCLUSION:

* Respiratory tract infection within the 4 weeks prior to Visit 0 Oral or systemic corticosteroid burst (for any indication) within the 4 weeks prior to Visit 0. One-time doses, such as intra-articular injections into a shoulder or knee joint, require a 4-week washout prior to Visit 0
* Significant concomitant medical illness, including (but not limited to) heart disease, cancer, uncontrolled diabetes, other chronic lung diseases
* Chronic renal failure (creatinine > 2.0) at Visit 0
* Positive urine pregnancy test at Visit 0 or at any time during the study
* Untreated sleep apnea
* Participation in an intervention study (including bronchoscopy) or use of investigative drugs within the past 30 days or plans to enroll in such a trial during the study
* Unable or unlikely to complete study assessments in the opinion of the Investigator
* Study intervention poses undue risk to patient in the opinion of the Investigator

Additional EXCLUSION Criteria for MRI

* Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements
* Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine, shoulder circumference >140 cm*.) *This measurement is not an absolute as it can vary based on weight distribution.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Percent trichrome or elastic or fiber staining between fixed and reversible airway segments in obese asthma groups (early onset, late onset) and non-asthma controls will be determined. | Up to 6 weeks
Percent neutrophils in peripheral blood in obese and lean asthmatics will be determined. | Up to 6 weeks
Percent eosinophils in peripheral blood in obese and lean asthmatics will be determined. | Up to 6 weeks
Percent change in 3-Nitrotyrosine production by airway epithelial cells harvested from obese and lean asthmatics and non-asthmatic obese controls will be determined. | Baseline, visit 1 (one week +/- 7 day), visit 2 (one week +/- 7 day), visit 3 (one week +/- 7 day)
Percent change in H202 production by airway epithelial cells harvested from obese and lean asthmatics and non-asthmatic obese controls will be determined. | Baseline, visit 1 (one week +/- 7 day), visit 2 (one week +/- 7 day), visit 3 (one week +/- 7 day)
Leptin stimulated human airway fibroblast invasiveness will be determined by counting mean numbers of invading fibroblasts in obese and lean asthmatics and non-asthmatic obese controls. | Up to 6 weeks
Percent change in intracellular ROS production by airway fibroblasts will be assessed using flow cytometry. | Baseline, visit 1 (one week +/- 7 day), visit 2 (one week +/- 7 day), visit 3 (one week +/- 7 day)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Que, MD, Principal Investigator — Duke
Locations (1):
- Duke Asthma Allergy and Airway Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No